CLINICAL TRIAL: NCT05701969
Title: Effect of Melatonin on Sleep Patterns of Resident Trainees During Night Float Shift
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Lauren Dunn, MD, Assistant Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSR210118
Record Dates: First submitted 2023-01-06; First posted 2023-01-27 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Sleep Disorders, Circadian Rhythm
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: a prospective double-blinded randomized control trial to investigate the effect of melatonin on sleep quantity and quality in resident physicians assigned to a night float system.
Masking Description: The research pharmacy will randomize the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin group (Experimental): These subjects will receive melatonin
  Interventions: Dietary Supplement: Melatonin
- Placebo group (Placebo Comparator): These subjects will receive placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Melatonin — Melatonin
  Arms: Melatonin group
Other: Placebo — Placebo control
  Arms: Placebo group

SUMMARY:
Anesthesiology residency requires extended and overnight shifts, which may negatively impact the quantity and quality of sleep.

Previous studies have investigated the effect of night float shift work on anesthesiology resident sleep and performance and demonstrated that total sleep quantity and time spent in deep and rapid eye movement (REM) sleep were significantly reduced during night float and did not return to baseline after 3 nights of recovery.

Melatonin is a hormone produced by the pineal gland, which regulates the circadian rhythm that governs sleep. Exogenous melatonin may be used as a sleep aid and is available over the counter in the United States. Melatonin is effective in realigning the circadian rhythm disorder caused by night shift work and increasing sleep duration; however, melatonin's effect on improving sleep in resident trainees has not been investigated. The investigators propose a prospective double-blinded randomized control trial to investigate the effect of melatonin on sleep quantity and quality in resident physicians assigned to a night float system.

DETAILED DESCRIPTION:
Residents in Post-Graduate Years 1-7 enrolled in residency programs with a night float system (anesthesiology, general surgery, obstetrics and gynecology, general medicine, and pediatrics) will be invited to participate in the study. A clinical study coordinator will assist in obtaining informed consent. After informed consent is obtained, participants will be randomized to receive either 3 mg melatonin or a matching placebo control. Medications will be prepared and randomization performed by the University of Virginia Pharmacy. Both participants and study coordinators will be blinded to the treatment group. Participants will be provided with a 12-day supply of medication at the start of the night float week. They will be instructed to take one capsule at least 20 minutes prior to going to bed at night or during the day after completing their night float shift. Subjects will be given a portable electroencephalography (EEG) monitor (ZMachine© Insight+ monitor (General Sleep Corporation, Euclid, OH))12 and will be shown how to apply the machine, monitor its functionality, and troubleshoot minor issues. They will be asked to wear the device for 2-3 nights of baseline sleep, 5-6 days of sleep during night float, and 3-4 nights of recovery following night float, for a total of 12 consecutive days. Baseline sleep data will serve as a control for each subject. EEG data collected will include: Light Sleep, Deep Sleep, REM, Arousals, Total Sleep Time, Sleep Efficiency, Latency to Persistent Sleep, Wake After Sleep Onset, Total Deep Sleep, Total REM Sleep, and Time Out of Bed. Data from two different night float periods separated by at least 2 weeks will be collected (one-week melatonin and one-week placebo in random order). Residents will also be asked to complete a daily questionnaire assessing daytime sleepiness (Epworth Sleepiness Scale) and the use of caffeine or other stimulants.

ELIGIBILITY:
Inclusion Criteria:

* Post-Graduate Year 1-5
* Current enrollment in anesthesiology, general surgery, obstetrics and gynecology, general medicine, or pediatrics residency at the Unversity of Virginia

Exclusion Criteria:

* Current use of sleep aids
* Diagnosed sleep disorder
* History of a pacemaker or other medical device.
* pregnant or breast-feeding females
* Bleeding disorders
* Depression
* High blood pressure
* Seizure disorders
* History of transplant on immunosuppression therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Total Sleep Time (TST) | 2 weeks
  Measured in hours and fraction of hours, with a portable electroencephalography monitor ZMachine© Insight+ monitor (General Sleep Corporation, Euclid, OH)

SECONDARY OUTCOMES:
Light Sleep | 2 weeks
  Measured in hours and fraction of hours, with a portable electroencephalography monitor ZMachine© Insight+ monitor (General Sleep Corporation, Euclid, OH)
Deep Sleep | 2 weeks
  Measured in hours and fraction of hours, with a portable electroencephalography monitor ZMachine© Insight+ monitor (General Sleep Corporation, Euclid, OH)
Rapid Eye Movement Sleep | 2 weeks
  Measured in hours and fraction of hours, with a portable electroencephalography monitor ZMachine© Insight+ monitor (General Sleep Corporation, Euclid, OH)
Latency to Persistent Sleep (LPS) | 2 weeks
  Measured in hours and fraction of hours, with a portable electroencephalography monitor ZMachine© Insight+ monitor (General Sleep Corporation, Euclid, OH)
Wake after Sleep Onset (WASO) | 2 weeks
  Measured in hours and fraction of hours, with a portable electroencephalography monitor ZMachine© Insight+ monitor (General Sleep Corporation, Euclid, OH)
Sleep Efficiency (SE) | 2 weeks
  monitor ZMachine© Insight+ monitor (General Sleep Corporation, Euclid, OH)

OTHER OUTCOMES:
Epworth Sleepiness Scale | 2 weeks
  Score 0-24 (Interpretation:
  0-7: Unlikely to be abnormally sleepy. 8-9: Average amount of daytime sleepiness.
  10-15: May be excessively sleepy depending on the situation. Consider seeking medical attention.
  16-24: Excessively sleepy, consider seeking medical attention.)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Dunn, MD PHD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No